CLINICAL TRIAL: NCT07250035
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Study of Jiedu Huayu Oral Prescription in the Treatment of Intracranial Hemorrhage Associated With Cerebral Amyloid Angiopathy
Brief Title: Jiedu Huayu Oral Prescription in the Treatment of Intracranial Hemorrhage Associated With Cerebral Amyloid Angiopathy
Acronym: CHN-CAA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Dongzhimen Hospital, Beijing (Other); The First Hospital of Jilin University (Other); Huairou Hospital of Traditional Chinese Medicine (Other); Weihai Wendeng District Central Hospital (Unknown); Nanyang First People's Hospital of Henan province (Unknown); Luohe Central Hospital (Unknown); Baofeng County People's Hospital (Unknown); Taoyuan County People's Hospital (Unknown); Qingdao Huangdao District Central Hospital (Unknown); Guantao County People's Hospital (Unknown); Lushan County Hospital of Traditional Chinese Medicine (Unknown); Yutian County Hospital of Traditional Chinese Medicine (Unknown); Xianghe County Hospital of Traditional Chinese Medicine (Unknown); Wuyuan County People's Hospital (Unknown); Jiyuan Hospital of Traditional Chinese Medicine (Unknown); Tonghua People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024ZD0522204
Record Dates: First submitted 2025-09-19; First posted 2025-11-25 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Amyloid Angiopathy
MeSH Terms: conditions — Cerebral Amyloid Angiopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo
- Experimental (Experimental)
  Interventions: Drug: Jiedu Huayu Oral Prescription

INTERVENTIONS:
Drug: Jiedu Huayu Oral Prescription — Jiedu Huayu Oral Prescription in the Treatment of Intracranial Hemorrhage Associated with Cerebral Amyloid Angiopathy
  Arms: Experimental
Drug: Placebo — A placebo similar to the Jiedu Huayu Oral Prescription
  Arms: Placebo Comparator

SUMMARY:
Cerebral hemorrhage, as a serious cerebrovascular disease, has the highest disability rate and mortality rate among all types of cerebrovascular diseases .It has brought a heavy burden to society. In China, the incidence of cerebral hemorrhage is much higher than that in Europe and America, and cerebral amyloid angiopathy (CAA) is one of the causes of primary cerebral hemorrhage However, there are relatively few related studies. Therefore, the research object of this subject focuses on patients with cerebral amyloid angiopathy, in view of their high recurrence rate of vascular events and the lack of treatment methods.It aims to deeply explore the detoxification and blood stasis removal treatment plan combining traditional Chinese and Western medicine to reduce vascular events for patients.

DETAILED DESCRIPTION:
Cerebral hemorrhage, as a serious cerebrovascular disease, has the highest disability rate and mortality rate among all types of cerebrovascular diseases .It has brought a heavy burden to society. In China, the incidence of cerebral hemorrhage is much higher than that in Europe and America, and cerebral amyloid angiopathy (CAA) is one of the causes of primary cerebral hemorrhage However, there are relatively few related studies. Therefore, the research object of this subject focuses on patients with cerebral amyloid angiopathy, in view of their high recurrence rate of vascular events and the lack of treatment methods.It aims to deeply explore the detoxification and blood stasis removal treatment plan combining traditional Chinese and Western medicine to reduce vascular events for patients. It is expected that this will be systematically evaluated through a multi-center, randomized, double-blind, mimic-controlled clinical trial.The effectiveness and safety of the protocol in reducing the incidence of vascular events were observed, and its impact on patients' cognitive function and neurological function was also examined. The research plan includes patients with CAA-related intracranial hemorrhage within 7 days of onset.The therapeutic effect was measured by indicators such as the proportion of vascular events in patients at different stages of the disease, including hematoma expansion rate and abnormal liver and kidney functions.The safety was evaluated based on the incidence rate, and the anti-inflammatory, antioxidant and other properties of traditional Chinese medicine prescriptions were explored with the aid of imaging and biological indicators.The mechanism for improving cerebrovascular function. It is expected that through this study, it will provide clinical treatment for patients with CAA-related intracranial hemorrhage.A brand-new and effective plan brings better prognosis to patients, reduces the medical burden on patients' families and lowers the social burden medical costs. At the same time, it will also provide important reference basis for subsequent related research and promote the integrated treatment of traditional Chinese and Western medicine.

ELIGIBILITY:
Inclusion Criteria:

* ① Possible or very likely CAA-ICH;

  * Within 7 days of onset; ③ Primary supratentorial intracerebral hemorrhage (bleeding volume ≤30ml);

    * GCS≥8 points;

      * NIHSS score ≤25 points; ⑥50≤age≤90 years old; ⑦ Gender is not limited; ⑧ The subject or their legal representative gives informed consent and signs the informed consent form.

Exclusion Criteria:

* Those who are known to be allergic to the components of the traditional Chinese medicine compound used in the experiment;

  * It is known that after treatment with vascular malformations, aneurysms, coagulation disorders, anticoagulant or antiplatelet drugs, Intracranial conditions caused by clear etiologies such as thrombolytic therapy, post-infarction hemorrhage transformation, hematological diseases, moyamoya disease, etc;

    * Patients with traumatic intracranial hemorrhage;

      * Patients with active peptic ulcers or other clear tendencies of rebleeding;

        * Patients with severe liver or kidney dysfunction (Note: Severe liver dysfunction is defined as ALT or AST being greater than.

          ⑥ Those who have received or are planning to undergo surgical treatment;

          ⑦ Those who suffer from other life-threatening serious diseases and have an expected survival time of less than six months;

          ⑧ Other conditions that significantly limit the evaluation of neurological function, prevent the completion of cranial magnetic resonance imaging, or affect the follow-up of patient;

          ⑨ Pregnant women, those planning to become pregnant or lactating women;

          ⑩Those who are currently participating in other interventional clinical trials.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Vascular events | 180 days after onset
  Incidence of vascular events, including hemorrhagic and ischemic vascular events.

SECONDARY OUTCOMES:
Incidence of Vascular Events at 30 Days | 30 days after onset
  Incidence of vascular events.
Incidence of Vascular Events at 90 Days | 90 days after onset
  Incidence of vascular events.
Incidence of Vascular Events at 1 Year | 1 year after onset
  Incidence of vascular events.
Changes in Neurocognitive Function | 180 days after onset
  Changes in neurocognitive function assessed by TICS-M, MMSE, and MOCA scales.
Neurological Function Recovery at 30 Days | 30 days after onset
  Neurological function recovery evaluated by mRS score.
Neurological Function Recovery at 90 Days | 90 days after onset
  Neurological function recovery evaluated by mRS score.
Neurological Function Recovery at 180 Days | 180 days after onset
  Neurological function recovery evaluated by mRS score.
Neurological Function Recovery at 1 Year | 1 year after onset
  Neurological function recovery evaluated by mRS score.
Changes in Quality of Life at 30 Days | 30 days after onset
  Changes in quality of life assessed by SF-36 and EQ-5D scales.
Changes in Quality of Life at 90 Days | 90 days after onset
  Changes in quality of life assessed by SF-36 and EQ-5D scales.
Changes in Quality of Life at 180 Days | 180 days after onset
  Changes in quality of life assessed by SF-36 and EQ-5D scales.
Changes in Quality of Life at 1 Year | 1 year after discharge
  Changes in quality of life assessed by SF-36 and EQ-5D scales.

OTHER OUTCOMES:
Safety Indicators at 7 Days | 7 days after onset
  Hematoma expansion rate in safety indicators (defined as a 33% increase in hematoma volume or an absolute increase of 6ml compared with the baseline CT hematoma volume).
Safety Indicators at 14 Days | 14 days after onset
  Hematoma expansion rate in safety indicators (using the same evaluation standard as that at 7 days after onset).
Safety Indicators during medication | During medication
  Incidence of newly developed severe liver and kidney function abnormalities in safety indicators.
Safety Indicators during entire study period | Entire study period
  Incidence of non-vascular death, adverse events/serious adverse events reported by researchers.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No